CLINICAL TRIAL: NCT06520748
Title: IMPACT OF COMPUTERIZED GLOVE ON FACILITATING HAND FUNCTION RECOVERY AND NEURAL PLASTICITY IN PATIENT WITH STROKE
Brief Title: IMPACT OF COMPUTERIZED GLOVE ON FACILITATING HAND FUNCTION RECOVERY AND NEURAL PLASTICITY IN STROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Alshimy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Alshimy, Lecturer of Physical Therapy for Neurology and it's Surgery, AlRyada University for Science & Technology
Organization: AlRyada University for Science & Technology (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004602
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Stroke; Hand recovery; Plasticity; Computerized glove
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): underwent a hand rehabilitation program using the computerized glove combined with the selected hand program
  Interventions: Other: Hand rehabilitation program using the computerized glove; Other: Selected hand program
- Control Group (Experimental): received only the selected hand program
  Interventions: Other: Selected hand program

INTERVENTIONS:
Other: Hand rehabilitation program using the computerized glove — The patient extended finger to reach from grey to green to red colour and heard the beep providing knowledge of result (KR), whereas the increase of range of finger extension reached every session provides knowledge of performance (KP). As the patient's performance improved, the range of their finger's movement will also be increased due to the augmented feedback provided to the patient and the therapist through the glove software
  Arms: Study Group
Other: Selected hand program — Distal key point of Bobath, approximation of affected arm, to control spasticity of wrist/ finger flexor (5 minutes). Dynamic splint to facilitate wrist and finger extension (10 repeat*5 sets). Passive range of motion exercise (10 repeat*5 sets) for each joint. Mud exercise (spherical, clyndrical , hook). Thera band exercises.

SUMMARY:
Hand impairment post-stroke is a common condition that contributes to disability around the world. An effective intervention is required to optimize functional outcomes in the rehabilitation of hand-in-stroke patients.

DETAILED DESCRIPTION:
Thirty male/female stroke patients in the sub-acute phase were randomly assigned in to the two groups (study and control) in sets of three. The study group (A) (n = 15) underwent a hand rehabilitation program using the computerized glove combined with the selected hand program. The control group (B) (n = 15) received only the selected hand program. The treatment schedules for 18 consecutive treatment sessions, three times per week.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age ranges from 45 to 65 years old with a minimum score of 24 points on the Mini Mental Test.
2. Duration of illness ranges from (6weeks to 6 months) after stroke onset.
3. first stroke.
4. Upper limb spasticity ranged from 1+ to 2 according to the Modified Ashworth Scale.
5. With a minimum 10° extension and/or flexion of the wrist or fingers, an ability to flex and extend the wrist joint five times continuously without losing active range of motion.

Exclusion Criteria: Patients with the following

1. apraxia or hemianopsia.
2. diabetic polyneuropathy.
3. Aphasia , cognitive deficits.
4. a previous disability in the upper limbs, tactile agnosia (stereognosis).
5. LT hemiplegia, Post Botox injection, recurrent stroke, and Posterior parietal lesion.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Quantitive Electro Encephalo Graphy | 6 weeks
  Used to assess Neuralplasticity (sleep Delta - Delta/Beta ratio )
Computerized glove software | 6 weeks
  Used to assess the Kinematic Data (Thumb, Index, Middle, ring, little, and average range of motion)
Action Research Arm Test | 6 weeks
  Used to assess Fine manual dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Al Ryada University for Science and Technology, Sadat, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No